CLINICAL TRIAL: NCT03569761
Title: A Randomized Trial of a Culturally-adapted Colorectal Cancer Screening Decision Aid Designed for American Indians
Brief Title: A Culturally-adapted Colorectal Cancer Screening Decision Aid Designed for American Indians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LCCC 1711
Record Dates: First submitted 2017-10-09; First posted 2018-06-26 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer screening; decision aids; American Indians
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The investigators will use a two-group randomized controlled trial to achieve our aims. Participants (n=120) will be randomized to view the AI culturally-adapted decision aid or an attention-control (i.e., food safety) video. The study flow diagram (Figure 2) indicates the recruitment, randomization, and assessment process.Our research to develop and evaluate the decision aid is approved by the Lumbee Tribal Council and the institutional review board (IRB) at the University of North Carolina at Chapel Hill.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision Aid Video Intervention (Experimental): Participants randomized to the intervention group will view the AI culturally-adapted CRC screening decision aid in a private room at a RHCC clinic. The video will be viewed on an electronic tablet or laptop computer.
  Interventions: Behavioral: Colorectal Cancer Screening Decision Aid
- Control (Active Comparator): Participants randomized to the control group will view an attention-control video about food safety in a private room at a RHCC clinic. The video will be viewed on an electronic tablet or laptop computer. The investigators chose the attention-control video so that the structure of the control arm mirrors the intervention arm. The food safety topic was chosen to provide information that is reasonably salient to the control arm participants but that would not be likely to affect encounters with healthcare providers.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Colorectal Cancer Screening Decision Aid — Information previously discussed in arm/group descriptions. There will be baseline, post-encounter, and 5-month follow-up assessments.
  Arms: Decision Aid Video Intervention
Behavioral: Control Group — Information previously discussed in arm/group descriptions. There will be baseline, post-encounter, and 5-month follow-up assessments. Information previously discussed in arm/group descriptions. There will be baseline, post-encounter, and 5-month follow-up assessments.
  Arms: Control

SUMMARY:
Experts note that in order to continue reducing the US cancer burden, it is critical that investigators "more completely apply discoveries in cancer prevention we have already made." Thus, it is important to research strategies that aim to improve application of effective colorectal cancer (CRC) prevention and screening tests among underserved populations like American Indians (AI).CRC is the 2nd leading cause of cancer death among AI; yet, one of the most preventable and treatable cancers when detected early. Increased use of recommended CRC screening tests among men and women ages 50-75 have contributed to nearly 50% declines in US CRC mortality since 1990. However, recent evidence indicates AI have not observed equitable improvements. The investigators propose to build upon our experience addressing CRC screening in underserved populations and strong partnerships with North Carolina tribal partners to gain new insight about a patient-centered, culturally appropriate strategy to increase AI CRC screening.

DETAILED DESCRIPTION:
Colorectal Cancer (CRC) Screening Options. CRC is a unique cancer due to the multiple screening options including stool-based (fecal occult blood testing (FOBT) and fecal immunochemical testing (FIT)), and direct visualization (colonoscopy) options. Healthcare providers tend to recommend colonoscopy, although evidence indicates that many patients, especially low-income and racial and ethnic minorities, prefer stool-based testing for a variety of reasons. In our formative work with North Carolina tribes, the investigators found evidence of low awareness of stool-based tests among American Indians (AI) and healthcare provider preferences to recommend colonoscopy. The US Preventive Services Task Force (USPSTF) guidelines indicate that evidence does not support favoring one CRC screening test above the others, and that recommendations should be based on patient preferences among the screening options. However, patient's general lack of knowledge of CRC screening modalities, literacy barriers to understanding differences between options, and other communication barriers in the healthcare setting (e.g., limited physician time) make this recommendation difficult to implement in practice without appropriate tools and support. Multimedia decision aids provide a practical solution to overcome communication challenges by providing patients information using easy-to-understand graphics and narratives designed to help them understand options, think through what is important to them, and engage with healthcare providers and family in the decision-making process.

CRC Screening Decision Aids. A recent systematic review and meta-analysis found evidence that average risk patients (aged 50 and over) exposed to CRC screening decisions aids showed greater increases in knowledge, were more likely to be interested in getting screened, and more likely to be screened. Most research on decision aids has been conduct with majority White populations; a few studies have focused on patients with low socioeconomic status. To our knowledge, no CRC screening decision aid studies have focused on AI populations.Our team has expertise in adapting CRC screening decision aids for underserved populations. The investigators have used a rigorous, community- and patient-engaged process to adapt a decision aid previously shown to be effective among majority White populations. The process retains effective elements of the existing version and refines content using messages and messengers that are culturally-sensitive (beyond peripheral packaging of graphics and visual content). A version the investigators adapted for low-income Hispanics significantly improved Hispanic patient's CRC screening knowledge, patient-provider communication, self-efficacy, and intent, and when combined with navigation, significantly improved completion of screening.

AI Barriers to CRC Screening. AI may benefit from decision aids; yet, CRC screening decision aids have not been developed or tested with AI populations. Several studies have found that AI have lower awareness and knowledge about CRC screening options and low perceived susceptibility of CRC than White populations. Many qualitative studies also indicate social and cultural barriers to CRC screening. For example, AIs indicate taboos related to speaking of illness or of certain body parts and fatalistic cultural beliefs influence their attitudes and intentions to obtain preventive medical services. In addition, a history of unethical healthcare practices and mistreatment of AI by the US government has led to issues of mistrust. Recent studies have found that AI report negative perceptions of medical providers and mistrust in healthcare institutions as barriers to obtaining CRC screening. Decision aids can address low awareness of options and improve attitudes and intentions for screening, especially if the content and the messengers of the information are adapted for sensitivity to relevant socio-cultural barriers (e.g., spiritual advisors who are credible to AI endorse screening). For this proposal, the investigators propose to test a novel culturally-adapted decision aid that aims to improve knowledge, attitudes and intentions to obtain CRC screening and uses messaging developed with our tribal community partners to overcome health literacy and socio-cultural barriers.

Conceptual Framework. Our decision aid is informed by the Theory of Planned Behavior and Cultural Identity Theory. The Theory of Planned Behavior posits that individual's attitudes (i.e., how one feels about a behavior and the potential outcomes of the behavior), norms (i.e., the amount of social pressure one feels to perform a behavior), and agency (i.e., the extent that one feels in control and able to perform a behavior) impacts their intentions to and subsequent performance of a behavior. The investigators also draw upon Cultural Identity Theory and posit that one's cultural identity and corresponding values underlie how one receives and interprets communicated messages and how one communicates with others about these messages. Our culturally-adapted decision aid uses messages that address AI-specific attitudes, norms, agency and communication concerns.

Preliminary Studies. With developmental funding from UNC's Lineberger Comprehensive Cancer Center, the investigators followed a rigorous process to adapt a general population version of a CRC screening decision aid for AI. From January to May of 2016, the investigators conducted six focus groups (n=74) with AI (ages 50-75) and interviews with healthcare providers (n=8) from three North Carolina tribal communities. The investigators explored perspectives about cultural, communication, and literacy barriers to CRC screening, and identified critical themes regarding AI cultural identity and socio-cultural values that influence CRC screening. The investigators and our tribal partners have operationalized the themes into adaptations of the existing general population decision aid. The decision aid provides information on stool-based and colonoscopy tests, the two types readily available in the community. The investigators are filming and making edits to the decision aid, which will be completed and ready for pilot testing by December 2016. Themes from AI focus groups and operationalized changes to a culturally-adapted CRC screening decision aid Operationalized Changes Healthcare mistrust - concern that inappropriate medical tests are recommended by providers Religious advisor to provide information and conveys trust in CRC screening options AI collectivism - stronger 'family' and community orientation toward health than individual focus New messages emphasize the benefit of CRC screening to one's family and community Privacy concerns- indication of difficulties and discomfort talking about CRC screening with family Vignette that models family communication around CRC screening Fear of cancer and screening - fear of cancer and screening process reduces motivation for screening AI CRC survivor to share experience of being screened and treated early

Methods A. Setting Our current research is centered in North Carolina tribal communities, primarily with the Lumbee Tribe of North Carolina, a state-recognized tribe that is located in Southeastern North Carolina. There are 62,306 Lumbee tribal members, the majority of whom (48,494) live in Robeson county. As with AI populations across the US, North Carolina AI have high rates of poverty and low educational attainment. One-third (33%) of AI in Robeson County are below the federal poverty level compared to 17% in North Carolina overall.45As a state-recognized tribe, Lumbee are not eligible for services through the federally-funded Indian Health Service,44 and many Lumbee tribal members use safety-net and federally qualified health centers such as the Robeson Health Care Corporation (RHCC), partner on this grant (see letter of support) to obtain health services.Robeson Health Care Corporation is a federally qualified health center with six clinics located in Robeson and neighboring counties. RHCC serves over 14,000 patients per year; 40% are AI. Nearly all, 95.6% of RHCC patients are at or below 200% of the federal poverty line. According to recent reports, 6,295 RHHC patients were not up-to-date with CRC screening following recommended guidelines.RHHC also has a long history of research collaboration on cancer screening projects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50-75
* Self-identify as AI (from any tribe)
* Are not up-to-date with recommended screening in accordance with USPSTF guidelines.

Exclusion Criteria:

* Patients who have a personal or family history of CRC or adenomatous polyps or inherited genetic conditions that increase CRC risk (familial adenomatous polyposis, Lynch syndrome, Turcot syndrome, Peutz-Jeghers syndrome, or MUTYH-associated polyposis)
* Unable to speak English
* Severe cognitive, visual, or hearing impairment that would prevent decision aid viewing.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
CRC screening intentions | Immediately after participant views their respective assigned video. Five (5) months following the encounter, a research assistant will call and administer a follow-up survey.
  Measure of screening intent from prior CRC screening decision aid studies and assessed using a single categorical item regarding intentions to get CRC screening with four response options.

SECONDARY OUTCOMES:
Knowledge | Immediately after participant views their respective assigned video. Five (5) months following the encounter, a research assistant will call and administer a follow-up survey.
  Assessed by a six-item index (based on decision aid content). Items include 1) the availability of more than one option for CRC screening; 2) the availability of a home screening test; 3) the recommended age to begin CRC screening; 4) FOBT screening test frequency; 5) the need for sedation (and companion driver) for colonoscopy procedure, and 6) the existence of a small but non-zero complication risk associated with having colonoscopy.
Attitudes | Immediately after participant views their respective assigned video. Five (5) months following the encounter, a research assistant will call and administer a follow-up survey.
  Assesses attitudes about how important items are for a participant's decision of whether or not to get CRC screening, including potential pros (e.g., having peace of mind after receiving clear findings) and cons (e.g., being worried or concerned that if you do the test you might find something wrong) with 4-point Likert-scale response options.
Perceived social norms | Immediately after participant views their respective assigned video. Five (5) months following the encounter, a research assistant will call and administer a follow-up survey.
  Assesses the participant's belief that family, friends, and doctors think he/she should be screened.
Personal agency | Immediately after participant views their respective assigned video. Five (5) months following the encounter, a research assistant will call and administer a follow-up survey.
  Assesses confidence to complete screening with 4-point Likert-scale response options (i.e., not at all confident, not very confident, confident, very confident).
CRC screening preferences | Immediately after participant views their respective assigned video. Five (5) months following the encounter, a research assistant will call and administer a follow-up survey.
  Measures screening preferences from prior studies.
Healthcare provider communication | Immediately after participant views their respective assigned video. Five (5) months following the encounter, a research assistant will call and administer a follow-up survey.
  Assessed with a participant-reported measure of having had a CRC screening discussion with a healthcare provider in the prior 5 months based on items used in a national survey.
Family and friend communication | Immediately after participant views their respective assigned video. Five (5) months following the encounter, a research assistant will call and administer a follow-up survey.
  Assessed using a measured adapted from a study on family communication about cancer screening. Participants asked to enumerate social network members and will be asked to identify members with whom they discussed CRC screening.
CRC screening completion | Immediately after participant views their respective assigned video. Five (5) months following the encounter, a research assistant will call and administer a follow-up survey.
  Dichotomous indicator of whether or not the participant completed any of the recommended CRC screening tests.

CONTACTS AND LOCATIONS:
Overall Officials: Leah Frerichs, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Robeson Health Care Corporation, Lumberton, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Frerichs L, Beasley C, Pevia K, Lowery J, Ferrari R, Bell R, Reuland D. Testing a Culturally Adapted Colorectal Cancer Screening Decision Aid Among American Indians: Results from a Pre-Post Trial. Health Equity. 2020 Apr 1;4(1):91-98. doi: 10.1089/heq.2019.0095. eCollection 2020. PMID 32258960